CLINICAL TRIAL: NCT03708003
Title: Ibrutinib lead-in Followed by Venetoclax Plus Ibrutinib in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia. A Multicenter, Open-label, Phase II Trial
Brief Title: Ibrutinib lead-in Followed by Venetoclax Plus Ibrutinib in Patients With RR CLL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The board decision has been made to conclude the trial ahead of schedule. The primary endpoint has been successfully achieved and published, and funding was secured to support these three years of followup.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 34/17
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Leukemia
Keywords: lymphocytic leukemia; relapsed/refractory chronic lymphocytic leukemia; Ibrutinib; venetoclax
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Leukemia, Lymphoid | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Intervention Model Description: A multicenter, single-arm, open-label, phase-II trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- venetoclax + ibrutinib (Experimental): Ibrutinib lead-in followed by venetoclax plus ibrutinib administered until cycle 31. The combination treatment will be continued as maintenance treatment or stopped depending on MRD-neg CR/CRi status.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Patients receive 6 cycles (cycle = 28 days) of ibrutinib monotherapy at the daily dose of 420 mg (3x 140 mg).
  Venetoclax is added on ibrutinib treatment starting from cycle 7 as weekly dose ramp-up (20 mg, C7 day 1-7; 50 mg, C7 day 8-14; 100 mg, C7 day 15-21; 200 mg, C7 day 22-28; 400 mg, C8-31 day 1-28).
  Venetoclax (400 mg d1-28) and ibrutinib (420 mg d1-28) continue until cycle 31. Depending on MRD-neg CR/CRi patients will continue the combination treatment (maintenance) or stop treatment (observation) up to 5 years after cycle 31.
  Other Names: Imbruvica
Drug: Venetoclax — Venetoclax is added on ibrutinib treatment starting from cycle 7 as weekly dose ramp-up (20 mg, C7 day 1-7; 50 mg, C7 day 8-14; 100 mg, C7 day 15-21; 200 mg, C7 day 22-28; 400 mg, C8-31 day 1-28).
  Venetoclax (400 mg d1-28) and ibrutinib (420 mg d1-28) continue until cycle 31. Depending on MRD-neg CR/CRi patients will continue the combination treatment (maintenance) or stop treatment (observation) up to 5 years after cycle 31.
  Other Names: Venclyxto

SUMMARY:
Venetoclax and ibrutinib have complementary activity in clearing the disease across anatomical compartments. By combining ibrutinib with venetoclax, cells can be mobilized from tissues into the bloodstream by ibrutinib and killed in the blood by venetoclax. Consistently, the venetoclax-ibrutinib combination can achieve undetectable minimal residual disease (MRD-neg) in a sizable proportion of patients. Gentle debulking obtained with a lead-in phase of ibrutinib monotherapy may allow starting venetoclax when the disease has been reshaped in a size that fits for low-risk of tumor lysis syndrome (TLS), a rare adverse event (AE) of venetoclax. MRD-guided treatment duration may allow patients achieving a negative status to gain drug-free intervals and less medicalization, and may avoid all the potential, and not yet completely known implications of continuous therapy on long-term safety, drug interactions, quality of life, compliance to treatment, and economic sustainability.

DETAILED DESCRIPTION:
Background:

The standard of care for treatment of patients with relapsed or refractory chronic lymphocytic leukemia (RR CLL) has substantially changed. Current standard for patients with a relapse later than 3 years from first-line therapy is a repetition with the first-line regimen used. This poses the risk of significant immunosuppression and infectious complications as well as a shorter event-free survival as expected for first-line treatment. Current standard for patients with refractory disease, early relapse or emerging TP53 defective clones, is a targeted treatment with ibrutinib, idelalisib + rituximab or venetoclax as continuous therapy until progression or toxicity.

Rationale:

Venetoclax and ibrutinib are both oral drugs whose tolerability when used in combination is not inferior to single agents. Venetoclax and ibrutinib have complementary activity in clearing the disease across anatomical compartments. Ibrutinib is more active in lymph nodes rather than blood where a small lymphocytosis might persist despite continuous treatment. Conversely, venetoclax appears to be more active in blood and bone marrow (BM) rather than lymph nodes. By combining ibrutinib with venetoclax, cells can be mobilized from tissues into the bloodstream by ibrutinib and killed in the blood by venetoclax. Consistently, the venetoclax-ibrutinib combination can achieve undetectable minimal residual disease (MRD-neg) in a sizable proportion of patients. Gentle debulking obtained with a lead-in phase of ibrutinib monotherapy may allow starting venetoclax when the disease has been reshaped in a size that fits for low-risk of tumor lysis syndrome (TLS), a rare adverse event (AE) of venetoclax. MRD-guided treatment duration may allow patients achieving a negative status to gain drug-free intervals and less medicalization, and may avoid all the potential, and not yet completely known implications of continuous therapy on long-term safety, drug interactions, quality of life, compliance to treatment, and economic sustainability.

The primary objective of the trial is to assess efficacy after 30 cycles of trial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration and prior to any trial specific procedures
* Cytologically and immunophenotypically confirmed relapsed/refractory CLL (irrespective of the 17p deletion and/or TP53 mutation status and the duration of remission from last prior therapy)
* Patients in need of systemic treatment as defined by international workshop on chronic lymphocytic leukemia (iwCLL) criteria (at least one of the following indications must be fulfilled):

  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia. Cut-off levels of Hb < 100 g/L or platelet counts of < 100x109/L
  * Massive (i.e., ≥ 6 cm below the left costal margin) or progressive or symptomatic splenomegaly
  * Massive nodes (i.e., ≥ 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy
  * Progressive lymphocytosis with an increase of ≥ 50% over a 2-month period, or lymphocyte doubling time of less than 6 months
  * Disease-related symptoms as defined by any of the following: (a) Unintentional weight loss ≥ 10% within the previous 6 months. (b) Significant fatigue (i.e., ECOG PS 2 or worse; cannot work or unable to perform usual activities). (c) Fevers ≥38.0° C for 2 or more weeks without evidence of infection. (d) Night sweats for ≥ 1 month without evidence of infection
* Age at least 18 years
* WHO performance status 0-2
* Hematological function:

  * Absolute neutrophil count (ANC) ≥ 1 x 109/L or ANC < 1 x 109/L, if attributable to the underlying CLL (growth factor support may be administered after screening)
  * Platelet count ≥ 30 x 109/L
* Hepatic function:

  * Bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN)
  * ALT and AST ≤ 3.0 x ULN
* Renal function: Creatinine clearance > 30 mL/min (calculated according to institutional standards or using Cockcroft-Gault formula
* Adequate coagulation parameters per local laboratory reference range as follows: activated partial thromboplastin time (aPTT) and international normalized ratio (INR) ≤ 1.5 × ULN
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and during the 30 days thereafter. A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential
* Men agree not to father a child during trial treatment and during 3 months thereafter
* Patient is able and willing to swallow trial drugs as whole tablet/capsule
* Patient is willing to participate in translational research

Exclusion Criteria:

Any potential patient who meets any of the following criteria has to be excluded from entering the trial.

* Transformation of CLL (i.e. Richter's transformation, prolymphocyctic leukemia)
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low-risk of recurrence and/or no late recurrence
* Prior treatment with venetoclax and/or ibrutinib
* Major surgery and any systemic anti-cancer treatment within 3 weeks prior to registration
* Steroid therapy for anti-neoplastic intent; strong and moderate CYP3A inhibitors; strong and moderate CYP3A inducers must be stopped at least 7 days prior to the first dose of trial drug (see http://medicine.iupui.edu/ and useful tools for examples)
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia on direct oral anticoagulants (DOAC), Aspirin or low molecular weight heparins (LMWH) but not on Vitamin K antagonist), significant QT-prolongation, uncontrolled hypertension
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to registration and known bleeding disorders (e.g., von Willebrand's disease or hemophilia)
* Patients with a history of confirmed progressive multifocal leukoencephalopathy (PML)
* Concomitant diseases that require anticoagulant therapy with warfarin or phenoprocoumon or other vitamin K antagonists. Patients being treated with factor Xa inhibitors (e.g. rivaroxaban, apixaban, edoxaban), direct thrombin inhibitors (e.g. dabigatran) LMWH, or anti-platelets agents (e.g. aspirin, clopidogrel) can be included, but must be properly informed about the potential risk of bleeding under treatment with ibrutinib
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Any uncontrolled active systemic infection requiring intravenous antimicrobial treatment
* Known history of human immunodeficiency virus (HIV) infection. Active hepatitis B infection (defined as the presence of detectable HBV DNA, HBe antigen or HBs antigen). Patients with serologic evidence of prior vaccination (HBsAg negative, anti-HBs antibody positive, anti-HBc antibody negative) are eligible. Patients who are HBsAg negative/HBsAb positive but HBcAb positive are eligible, provided HBV DNA is negative. Active hepatitis C, defined by the detectable hepatitis C ribonucleic acid (RNA) in plasma by polymerase chain reaction (PCR)
* Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy with > 20mg daily of prednisone dose or equivalent
* Known hypersensitivity to trial drugs or to any component of the trial drugs
* Known allergy to both xanthine oxidase inhibitors and rasburicase
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and/or would make the patient inappropriate for enrollment into this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
MRD-neg CR/CRi at end of cycle 30 | after 840 days (1 cycle = 28 days)
  The MRD-neg (Undetectable Minimal residual disease) Complete remission/Complete remission with incomplete marrow recovery CR/CRi rate is defined as the proportion of patients having achieved:
  * CR/CRi, according to the iwCLL (International workshop on chronic lymphocytic leukemia) guidelines (2018), and
  * MRD-neg in bone marrow BM, measured by flow cytometry with a quantitative lower limit of at least < 10-4. MRD status will be considered as negative if the proportion of malignant cells is < 10-4.
  Patients without any response or MRD BM assessment at end of cycle 30 (+/- 14 days) will be counted as non-responders (failures for the primary endpoint).

SECONDARY OUTCOMES:
ORR at end of cycle 30 | after 840 days (1 cycle = 28 days)
  The ORR (Overall response rate) is defined as the proportion of patients having achieved a CR/CRi or PR according to the iwCLL guidelines (2018) and will be evaluated at end of cycle 30 (+/- 14 days). Patients without any response assessment at end of cycle 30 (+/- 14 days) will be counted as non-responders.
CR/CRi rate at end of cycle 30 | after 840 days (1 cycle = 28 days)
  The CR/CRi rate (Complete remission/Complete remission with incomplete marrow recovery) is defined as the proportion of patients having achieved a CR/CRi according to the iwCLL guidelines (2018) and will be evaluated at end of cycle 30 (+/- 14 days). Patients without any response assessment at end of cycle 30 (+/- 14 days) will be counted as non-responders.
CR/CRi rate based on best response | Day 1 of cycle 7, 13, 19, 25 and 31 (1 cycle = 28 days)
  The CR/CRi rate based on best response is defined as the proportion of patients having achieved a CR/CRi according to the iwCLL guidelines (2018) as best response during trial therapy including maintenance. Patients without any post-baseline response assessment will be counted as non-responders.
MRD-neg rate | Day 1 of cycle 7, 13, 19, 25 and 31 (1 cycle = 28 days)
  The MRD-neg rate is defined as the proportion of patients having achieved MRD-neg at any time during trial therapy including maintenance. Patients without any post-baseline MRD assessment will be counted as MRD positive patients. As MRD status will be assessed from PB or BM, both PB MRD-neg rate and BM MRD-neg rate will be calculated.
Progression-free survival (PFS) | Day 169, 337, 505, 673, 841, yearly up to five years, end of trial treatment plus unscheduled (if progression is suspected)
  PFS is defined as the time from registration until progression according the iwCLL criteria or death from any cause, whichever occurs first. Patients not having an event at the time of analysis as well as patients starting a new antileukemic therapy in the absence of an event will be censored at the date of their last tumor assessment showing nonprogression before starting a new anti-leukemic treatment, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Rossi, MD, Study Chair — Institute of Southern Switzerland IOSI, Bellinzona
Locations (11):
- Switzerland (11):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - IOSI - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Liestal, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Münsterlingen, Münsterlingen
  - Spital STS AG Thun, Thun
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich, Zurich

REFERENCES:
- [Derived] Condoluci A, Romano I, Dietrich D, Pini K, Stussi G, Muller G, Cantoni N, Cathomas R, Mey U, Widmer A, Zenz T, Gregor M, Heim D, Andres M, Benz R, Rossi D. Ibrutinib lead-in followed by venetoclax plus ibrutinib for relapsed/refractory chronic lymphocytic leukemia: the SAKK 34/17 trial. Blood. 2025 May 29;145(22):2587-2598. doi: 10.1182/blood.2024026879. PMID 40009495